CLINICAL TRIAL: NCT05495919
Title: The Effectiveness of Different Teaching Models in Nursing Education in the Pandemic: Randomized Controlled Experimental Research
Brief Title: Nursing Education in the Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202151
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Anxiety; Satisfaction
Keywords: Pandemic; nursing education; model use in education; anxiety; satisfaction with education
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): No intervention was performed to reduce anxiety in the control group
  Interventions: Other: Control
- video interaction group (Experimental): Before the training, the students took videos and during the lesson, the videos were evaluated and feedback was given.
  Interventions: Other: video interaction
- Flipped Training (Experimental): Before the training, educational materials were given to the students, and they were discussed with the students in the lesson.
  Interventions: Other: flipped training

INTERVENTIONS:
Other: Control — No intervention was perfomed to reduce anxiety in control group
  Arms: Control Group
Other: video interaction — Before the training, educational materials were given to the students, and they were discussed with the students in the lesson.
  Arms: video interaction group
Other: flipped training — Before the training, the students took videos and during the lesson, the videos were evaluated and feedback was given.
  Arms: Flipped Training

SUMMARY:
One of the areas that has been badly affected during the current pandemic process is education. There is a need to use innovative teaching models in order to increase the efficiency of online education, which the pandemic has made compulsory, to involve the student in the lesson interactively and to increase the success level of the lesson. This study was planned as a randomized controlled experimental study in order to evaluate the effectiveness of different teaching models in nursing education during the pandemic.

DETAILED DESCRIPTION:
Material and method of the research:

Type of Study: The study was designed as randomized controlled experimental type.

Research Hypotheses Hypothesis 1 (H1): Nursing students who receive education using video interaction and flipped teaching model have less anxiety than students who receive education with the classical teaching model.

Hypothesis 2 (H2): The satisfaction level of nursing students who receive education using video interaction and flipped teaching model is higher than the students who receive education with the classical teaching model.

Population and Sample of the Study: The universe of the research; In the 2020-2021 academic year, 200 students will be enrolled in the Fundamentals of Nursing course in the Nursing Department of a state and a foundation university in June 2021 in the spring semester. Power analysis (NCSS-PASS Statistical package) was carried out to determine the number of students who will form the research sample. In order to carry out a study with P ≤ 0.1 levels of this analysis, it was decided to have 90 samples. Students in the sample group will be determined by randomization by the researcher. The students to be included in the study were made by randomization and selection method from the random numbers table. For randomization, a randomization table will be created by using the http://stattrek.com/statistics/random-number-generator.aspx site. As a result, the sample of the research; The purpose of the study will be explained and a total of 90 students who have been given permission to participate in the research after the information and who meet the sampling criteria of the research will be formed. The sampling criteria of the study; To be 18 years or older, not to be graduated from Health Vocational High School, to be registered for the first time in the Nursing Fundamentals course, to fully participate in the interventions to be applied in the study and to volunteer to participate in the study.

Data Collection Tools: Data were collected using the "Structured Student Introduction Form", "Static and Trait Anxiety Inventory" and "Satisfaction with Educational Methods Questionnaire".

Analysis of Data: Data were analyzed with SPSS 25 Package program.

ELIGIBILITY:
Inclusion Criteria:

Nursing Students,

* be between the ages of 18-25,
* not being a Health Vocational High School graduate,
* to be enrolled in the Nursing Fundamentals course for the first time,
* participating fully in the initiatives to be implemented in the study
* volunteering to participate in the study.

Exclusion Criteria:

Nursing Students,

* not between the ages of 18-25,
* health Vocational High School graduate,
* not being enrolled in the Nursing Fundamentals course for the first time,
* failure to fully participate in the initiatives to be implemented in the study
* not being willing to participate in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety Severity | 2 Months
  Students were informed about the State-Trait Anxiety inventory.

SECONDARY OUTCOMES:
Satisfaction Severity | 2 Months
  Students were informed about the education satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, PhD RN, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Beykent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leighton K, Kardong-Edgren S, McNelis AM, Foisy-Doll C, Sullo E. Traditional Clinical Outcomes in Prelicensure Nursing Education: An Empty Systematic Review. J Nurs Educ. 2021 Mar 1;60(3):136-142. doi: 10.3928/01484834-20210222-03. PMID 33657230
- [Result] Huang TH, Liu F, Chen LC, Tsai CC. The acceptance and impact of Google Classroom integrating into a clinical pathology course for nursing students: A technology acceptance model approach. PLoS One. 2021 Mar 5;16(3):e0247819. doi: 10.1371/journal.pone.0247819. eCollection 2021. PMID 33667246